CLINICAL TRIAL: NCT05763199
Title: Feasibility Pilot Study of a Standardized Extract of Cultured Lentinula Edodes Mycelia (AHCC®) on Quality of Life for Ovarian Cancer Patients on Adjuvant Chemotherapy
Brief Title: Standardized Extract of Cultured Lentinula Edodes Mycelia (AHCC®) in Ovarian Cancer Patients on Adjuvant Chemotherapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Amino Up Chemicals Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Hui Amy Chen, Assistant Professor, University of California, Davis
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UCDCC#302
Record Dates: First submitted 2023-01-27; First posted 2023-03-10 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Ovarian Epithelial Carcinoma; Fallopian Tube Carcinoma; Peritoneal Carcinoma
Keywords: AHCC; Standardized extract of cultured Lentinula edodes mycelia
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms | interventions — Drug Therapy; Platinum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standardized Extract of Cultured Lentinula Edodes Mycelia (AHCC®) (Experimental): AHCC 3g PO Daily
  Interventions: Dietary Supplement: AHCC; Drug: Chemotherapy
- Placebo (Placebo Comparator): Placebo PO Daily
  Interventions: Drug: Chemotherapy; Other: Placebo

INTERVENTIONS:
Dietary Supplement: AHCC — AHCC is the cultured mycelia of Lentinula edodes mushrooms from the Basidiomycetes family.
  Other Names: A standardized extract of cultured Lentinula edodes mycelia
  Arms: Standardized Extract of Cultured Lentinula Edodes Mycelia (AHCC®)
Drug: Chemotherapy — Chemotherapy will be administered per standard of care.
  Other Names: Platinum and taxane chemotherapy
Other: Placebo — Dextrin
  Arms: Placebo

SUMMARY:
This is a pilot phase, randomized, double-blinded feasibility pilot study of AHCC in participants with ovarian cancer.

DETAILED DESCRIPTION:
This is a pilot phase, randomized, double-blinded feasibility pilot study of AHCC in participants with ovarian cancer. 20 women who plan to undergo adjuvant chemotherapy for ovarian cancer at the University of California (UC) Davis Health Comprehensive Cancer Center will be enrolled and randomized 1:1 to receive AHCC (3 grams by mouth daily) or placebo during standard of care chemotherapy. HRQOL and adverse events will be assessed at baseline and during chemotherapy. The hypothesis is that a randomized controlled trial of AHCC supplementation for ovarian cancer patients on adjuvant chemotherapy is feasible.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed epithelial ovarian, fallopian tube or peritoneal carcinoma

   * High-grade or low-grade serous, mucinous, endometrioid, clear cell, mixed or other histologies allowed
2. Clinical stage I-IV at diagnosis
3. Treatment decision to include standard-of-care adjuvant chemotherapy after primary or interval debulking surgery, or initial staging surgery. Chemotherapy should include a platinum and a taxane doublet.

   * Neoadjuvant chemotherapy is allowed (no washout period will be required)
   * Any combination of platinum and taxane doublet is allowed (i.e., carboplatin, cisplatin, paclitaxel, or docetaxel)
   * Different schedules of platinum and taxane doublet are allowed (i.e., every 21 days, dose-dense or weekly)
   * Bevacizumab is allowed
4. Age greater than or equal to 18 years of age
5. English or Spanish-speaking individuals
6. Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2 (Karnofsky greater than or equal to 60%)
7. Organ and bone marrow function defined by:

   * Leukocytes greater than or equal to 2,500/µL
   * Absolute neutrophil count greater than or equal to 1,000/µL
   * Platelets greater than or equal to 75,000/µL
   * Hemoglobin greater than or equal to 8 g/dL
   * Total bilirubin less than or equal to 1.5 × institutional upper limit of normal (ULN) (however, patients with known Gilbert disease who have serum bilirubin level less than or equal to 3 x ULN may be enrolled)
   * Aspartate aminotransferase (AST)/ alanine transaminase (ALT) less than or equal to 3 × ULN (AST and/or ALT less than or equal to 5 x ULN for patients with liver involvement)
   * Alkaline phosphatase less than or equal to 2.5 × ULN (less than or equal to 5 x ULN for patients with documented liver involvement or bone metastases)
   * Creatinine clearance or glomerular filtration rate (GFR) greater than or equal to 30 mL/min by Cockcroft-Gault or 30 mL/min/1.73m2
8. Individuals of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) for the duration of study participation (including dosing interruptions) and for at least 5 months (150 days) after the last dose of study agent or the duration specified in the United Surgical Partners International (USPI) for any of the agents used in the adjuvant standard-of-care regimen, whichever is longest. Patients must agree to refrain from egg donation during this timeframe.
9. Ability to understand and the willingness to sign a written informed consent document
10. Patients with known human immunodeficiency virus (HIV) are allowed in the study, but HIV-positive patients must have:

    * A stable regimen of highly active anti-retroviral therapy (HAART)
    * No requirement for concurrent antibiotics or antifungal agents for the prevention of opportunistic infections
    * A cluster of differentiation 4 (CD4) count above 250 cells/µL and an undetectable HIV viral load on standard polymerase chain reaction (PCR)-based tests within the last year.

Exclusion Criteria:

1. History of allergic reactions to mushrooms
2. History of allergic reaction to dextrin
3. History of allergic reaction to rapeseed oil
4. History of allergic reaction to corn
5. Consumption of other supplements derived from mushrooms or basidiomycetes

   * Consumption of whole mushrooms through diet is acceptable
   * Consumption of a blend with unknown/ unclear mushrooms or basidiomycetes contents, then it is ok to include participant
6. Current or prior (within 3 months of enrollment) use of immunosuppressive medications (including, but not limited to, prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor (anti-TNF) agents). The following are exceptions to this criterion:

   * Intranasal, inhaled, topical or local steroid injections (e.g., intra-articular injection); steroids as premedication for hypersensitivity reactions; systemic corticosteroid at physiologic doses not to exceed 10 mg/day of prednisone or equivalent may be enrolled.
   * Patients who have received acute, low-dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) may be enrolled.
   * The use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension or adrenocortical insufficiency is allowed.
7. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would interfere with patient safety or limit compliance with study requirements.
8. Inability to swallow experimental agent or placebo
9. History of gastrectomy or other malabsorption syndromes
10. Subjects who are pregnant or breast-feeding
11. Any condition that would prohibit the understanding or rendering of informed consent
12. Any medical condition that in the opinion of the investigator would interfere with the patient's safety or compliance while on trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants consent and randomized to taking AHCC or placebo during adjuvant chemotherapy compared to to total number of ovarian cancer patients eligible for the trial following prescreening and participation invitation. | Study activation to randomization of 20th participant
Time required to randomize 20 participants | Study activation to randomization of 20th participant.
Proportion of participants that complete study treatment | First dose through Cycle 3-6 post adjuvant chemotherapy; each cycle is 3 weeks

SECONDARY OUTCOMES:
Proportion of participants that adhere to taking study treatment | First dose through Cycle 3-6 post adjuvant chemotherapy; each cycle is 3 weeks
Adherence to taking study treatment for each participant | First dose through Cycle 3-6 post adjuvant chemotherapy; each cycle is 3 weeks
Proportion of participants that adhere to completing the Functional Assessment of Cancer Therapy - Ovarian (FACT-O) | Baseline through 30d post last dose
  All health-related quality of life assessments use a 5 point Likert-type scale and is scored based on a manual scoring template, some items are reverse scored; the higher the score, the better the quality of life.
Proportion of participants that adhere to completing the Functional Assessment of Cancer Therapy/ Gynecologic Oncology Group - Neurotoxicity (FACT/ GOG-NTX) | Baseline through 30d post last dose
  All health-related quality of life assessments use a 5 point Likert-type scale and is scored based on a manual scoring template, some items are reverse scored; the higher the score, the better the quality of life.
Proportion of participants that adhere to completing the Functional Assessment of Cancer Therapy - Endocrine Symptoms (FACT-ES) | Baseline through 30d post last dose
  All health-related quality of life assessments use a 5 point Likert-type scale and is scored based on a manual scoring template, some items are reverse scored; the higher the score, the better the quality of life.
Participant experience self-reported in the acceptability questionnaire compared to self-reported anticipated acceptability | Baseline and at end of treatment (about 9-18 weeks post adjuvant chemotherapy)
  The acceptability questionnaire measures the following ordinal data listed in order of most acceptable to least acceptable: strongly agree, agree, neutral, disagree, and strongly disagree.

CONTACTS AND LOCATIONS:
Overall Officials: Hui Chen, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Comprehensive Cancer Center, Sacramento, California, United States